CLINICAL TRIAL: NCT01997333
Title: A Randomized Multicenter Pivotal Study of CDX-011 (CR011-vcMMAE)in Patients With Metastatic, gpNMB Over-Expressing, Triple Negative Breast Cancer (The METRIC Study)
Brief Title: Study of Glembatumumab Vedotin (CDX-011) in Patients With Metastatic, gpNMB Over-Expressing, Triple Negative Breast Cancer
Acronym: METRIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX011-04
Expanded Access: NCT03067935 (No longer available)
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Metastatic gpNMB Over-expressing Triple Negative Breast Cancer
Keywords: Metastatic Breast Cancer; Locally advanced breast cancer; Breast cancer; Triple negative; Estrogen; Progesterone; HER2 receptors; Targeted treatment for breast cancer; Antibody-drug-conjugate; Breast Neoplasms; CDX-011; gpNMB; METRIC; Glembatumumab vedotin; Triple Negative Breast Cancer; TNBC
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — glembatumumab vedotin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine (Active Comparator): Capecitabine will be administered on Days 1 through 14 of each 21 day cycle.
  Interventions: Drug: Capecitabine
- Drug: CDX-011 (Experimental): CDX-011 administered as an intravenous infusion on Day 1 of each 21 day cycle.
  Interventions: Drug: CDX-011

INTERVENTIONS:
Drug: CDX-011
  Arms: Drug: CDX-011
Drug: Capecitabine
  Arms: Capecitabine

SUMMARY:
The main purpose of this study is to see whether CDX-011 (glembatumumab vedotin, an antibody-drug conjugate) is effective in treating patients who have advanced Triple-Negative Breast Cancer (TNBC), and whose tumor cells make a protein called glycoprotein NMB (gpNMB), which CDX-011 binds to. The study will also further characterize the safety of CDX-011 treatment in this patient population.

DETAILED DESCRIPTION:
CDX-011 consists of an antibody attached to a drug, monomethyl auristatin E (MMAE), that can kill cancer cells. The antibody delivers the drug to cancer cells by attaching to a protein called glycoprotein NMB (gpNMB) that is expressed on the cancer cell. The MMAE is then released inside of the cell, where it interferes with cell growth and may lead to cell death.

This study will examine the efficacy and safety of CDX-011 in patients with advanced TNBC that makes the gpNMB protein. The effect of CDX-011 will be compared to treatment with capecitabine.

Eligible patients who enroll in the study will be randomly assigned (by chance) to receive treatment with CDX-011 or with capecitabine. For every three patients enrolled, two will receive CDX-011 and one will receive treatment with capecitabine. All patients enrolled in the study will be closely monitored to determine if their cancer is responding to treatment and for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet all of the following conditions to be eligible for the study:

1. Diagnosed with metastatic (i.e., cancer that has spread) TNBC

   * minimal or no expression of estrogen and progesterone receptors (ER/PR) <10% of cells positive by immunohistochemistry
   * HER 2 staining 0 or 1+ by IHC or copy number <4.0 signals/cell
2. Documented progression of disease based on radiographic, clinical or pathologic assessment during or subsequent to the last anticancer regimen received.
3. Breast cancer tumor confirmed to express gpNMB. This will be determined by submitting a tissue sample from the advanced (locally advanced/recurrent or metastatic) disease setting to a central laboratory for analysis.
4. Received no more than two prior chemotherapy treatments for advanced (locally advanced/recurrent or metastatic) breast cancer.
5. Prior chemotherapy treatment must have contained an anthracycline (e.g. doxorubicin or Doxil) if clinically indicated and a taxane (eg: Taxol).
6. ECOG performance status of 0 - 1.
7. Adequate bone marrow, liver and renal function.

Exclusion:

Among other criteria, patients who meet any of the following conditions are NOT eligible for the study:

1. Progression/recurrence of breast cancer during or within 3 months of completion of neoadjuvant or adjuvant chemotherapy.
2. Ongoing neuropathy or other chemotherapy or radiation-related toxicities that are moderate (Grade 2) or worse in severity.
3. Known brain metastases, unless previously treated and asymptomatic for 2 months and not progressive in size or number for 2 months.
4. Significant cardiovascular disease.
5. Previously received capecitabine and discontinued due to progression or intolerance; previously received CDX-011 or other MMAE containing agents.
6. Active systemic infection requiring treatment. Infection controlled by oral therapy will not be exclusionary.
7. Chronic use of systemic corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2013-11; Primary Completion 2017-11-30 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (140):
- United States (71):
  - Alabama Oncology, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Insititute, Mobile, Alabama
  - Arizona Cancer Research Alliance, Glendale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Compassionate Care Research Group, Fountain Valley, California
  - St. Jude Heritage Medical Group, Fullerton, California
  - USC Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Pacific Cancer Care, Salinas, California
  - University of California San Francisco, San Francisco, California
  - Kaiser Permaente, Vallejo, California
  - Wellness Hematology Oncology, West Hills, California
  - University of Miami Miller School of Medicine, Deerfield Beach, Florida
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Peachtree Hematology Oncology Consultants, PC, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Georgia Cancer Specialists Clinic, Atlanta, Georgia
  - Northwest Georgia Oncology Centers P.C., Marietta, Georgia
  - Summit Cancer Care, PC-Savannah, Savannah, Georgia
  - University of Chicago, Chicago, Illinois
  - Ingalis Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare, Peoria, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Hematology and Oncology Specialists, Marrero, Louisiana
  - Louisiana State University Health New Orleans, New Orleans, Louisiana
  - Oschner Medical Center, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Virginia Piper Cancer Center, Minneapolis, Minnesota
  - HCA Midwest Health, Kansas City, Missouri
  - Washington University Dept of Oncology, St Louis, Missouri
  - St John's Mercy Medical Center, St Louis, Missouri
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Clinical Research Alliance, Inc., Lake Success, New York
  - ProHEALTH Care Associates, Lake Success, New York
  - Beth Isreal Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Novant Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic-Taussig Cancer Institute-R35, Cleveland, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Mercy Clinic of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Beaverton, Oregon
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Charleston Hematology Oncology Associates (CHOA), Charleston, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Center for Biomedical Research, LLC, Knoxville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Oncology Hematology Consultants PA, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (9):
  - St. Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Western Hospital, Footscray, Victoria
  - Joint Ludwig-Austin Dept of Medical Oncology, Heidelberg, Victoria
  - Epworth Health Care, Richmond, Victoria
- Belgium (5):
  - GasthuisZusters Antwerpen, Wilrijk, Antwerpen
  - Grand Hopital de Charleroi asbl, Charleroi, Hainaut
  - UZ Leuven, Leuven, Vlaams Brabant
  - Institute Jules Bordet, Brussels
  - Clinique Edith Cavell, Brussels Capital Region
- Canada (5):
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Sunnybrook Health Sciences Centre Odette Cancer Center, Toronto, Ontario
  - St. MIchael's Hospital, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - Universite de Montreal-Hopital Du Sacre-Coeur De Montreal, Montreal, Quebec
- France (10):
  - Centre Antoine Lacassagne Centre Régional de Lutte Contre Le Cancer, Nice, Alpes-Maritimes
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon, Rhône
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans, Sarthe
  - Institut Sainte Catherine, Avignon
  - Centre Oscar Lambret, Lille
  - Hôpital de La Croix Rousse, Lyon
  - Centre Hospitalier de Mont de Marson - Hôpital Layné, Mont-de-Marsan
  - Institut Curie, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - Centre Hospitalier Prive Saint-Gregoire, Saint-Grégoire
- Germany (11):
  - Klinikum Essingen GmbH, Esslingen am Neckar, Baden-Wurttemberg
  - Helios Klinikum Berlin Buch, Berlin
  - Kliniken der Stadt Koeln gGmbH - Krankenhaus Holweide, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universität Des Saarlandes, Homberg (Efze)
  - Rotkreuzklinikum München, Munich
  - Universitätsklinikum Münster, Münster
  - Hämatologisch-Onkologische Schwerpunktpraxis, Troisdorf
- Italy (10):
  - Istituto Scientifico romagnolo Per Lo Studio E La Cura Del Tumori IRST, Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Azienda Ospedaliera Fatebenefratelli e Oftaimico, Milan, Lombardy
  - Istituto Nazionale Dei Tumori, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Centro Di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Azienda Ospedaliera Citta della Salute e della Scienza de Torino, Torino
- Spain (11):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellón
  - Hospital Universitario Ramon y Cajal, Madrid, Communidad Delaware
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - MD Anderson Cancer Center Madrid-Espana, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (8):
  - Barts Health NHS Trust, London, City of London
  - Derriford Hospital, Plymouth, Devon
  - Royal Sussex County Hospital, Brighton, East Sussex
  - Beatson West of Scotland Cancer Centre, Glasgow, Glasgow City
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - University College London, London, London, City of
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Sarah Cannon Research Institute UK, City of London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1531 patients screened to randomize 327 patients. Most common reasons for screen failure were tumor tissue inadequate/gpNMB negative (697), failure to meet other eligibility (256) and refused to participate (77).
Groups:
- Capecitabine: Capecitabine administered on Days 1 through 14 of each 21 day cycle until disease progression, discontinuation due to toxicity, withdrawal of consent, or end of study.
- CDX-011: CDX-011 administered on Day 1 of each 21 day cycle until disease progression, discontinuation due to toxicity, withdrawal of consent, or end of study.
Period: Randomization and Treatment
Arm/Group | Capecitabine | CDX-011
Started | 109 | 218
Completed (Completed = continuing to receive treatment at time of analysis) | 6 | 15
Not Completed | 103 | 203
Not completed — Disease Progression | 70 | 159
Not completed — Adverse Event | 10 | 32
Not completed — Physician Decision | 0 | 4
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Did not receive treatment | 17 | 5
Period: Survival Follow up
Arm/Group | Capecitabine | CDX-011
Started (Only patients who received treatment are included in survival follow up.) | 92 | 213
Completed | 76 | 199
Not Completed | 16 | 14
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Lost to Follow-up | 0 | 6
Not completed — Various | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capecitabine | CDX-011 | Total
Number analyzed (Participants) | 109 | 218 | 327
Age, Continuous [Median (Full Range); unit: years] | 55 [31 to 85] | 55 [28 to 85] | 55 [28 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 218 | 327
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 99 | 191 | 290
  Unknown or Not Reported | 5 | 16 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 9 | 20 | 29
  White | 91 | 176 | 267
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 16 | 23
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 5 | 12
  Belgium | 2 | 6 | 8
  United States | 72 | 143 | 215
  Italy | 6 | 7 | 13
  United Kingdom | 5 | 6 | 11
  Australia | 3 | 15 | 18
  France | 4 | 14 | 18
  Germany | 5 | 9 | 14
  Spain | 5 | 13 | 18
Number of prior relapses in advanced stage [Number; unit: participants]
  0 | 21 | 45 | 66
  1 | 58 | 122 | 180
  2 | 24 | 42 | 66
  3 | 6 | 9 | 15
Number of cytotoxic regimens in advanced stage [Median (Full Range); unit: cytotoxic regimen] | 1 [0 to 4] | 1 [0 to 3] | 1 [0 to 4]
Prior Taxane Use [Count of Participants; unit: Participants] | 108 | 218 | 326
Prior Anthracycline Use [Count of Participants; unit: Participants] | 95 | 185 | 280
Progression Free Interval post last Taxane [Count of Participants; unit: Participants]
  less than or equal to 6 months | 51 | 112 | 163
  greater than 6 months | 58 | 106 | 164

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the earlier of disease progression or death due to any cause. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or progression in a non-target lesion, or the appearance of new lesions. The primary analysis of PFS was based on PFS events determined retrospectively by the central independent review committee, blinded to treatment assignment and investigator assessments according to RECIST 1.1 criteria.
Time Frame: Evaluated every 6 - 9 weeks following treatment initiation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine | CDX-011
Number analyzed (Participants) | 109 | 218
months | 2.8 [1.6 to 3.2] | 2.9 [2.8 to 3.5]
Statistical Analysis 1: Comparison: Capecitabine vs CDX-011; Test type: Superiority; p = 0.761, Log Rank; Stratified log rank test

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients who achieve best overall response of complete or partial response. The analysis of ORR was based on ORR events determined retrospectively by the central independent review committee, blinded to treatment assignment and investigator assessments according to RECIST 1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Complete Response (CR) = Disappearance of all target lesions and non-target lesions, Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions with no progression in non-target lesions and no new lesions.
Time Frame: Evaluated every 6 - 9 weeks following treatment initiation
Population: Patients with measurable disease.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine | CDX-011
Number analyzed (Participants) | 100 | 179
percentage of participants | 21 [14 to 30] | 26 [20 to 33]
Statistical Analysis 1: Comparison: Capecitabine vs CDX-011; Test type: Superiority; p = 0.264, Cochran-Mantel-Haenszel; Adjusted for stratification factors

3. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) is the number of months from the time criteria are first met for either CR or PR, until the first date that PD is objectively documented. The analysis of DOR was determined retrospectively by the central independent review committee,blinded to treatment assignment and investigator assessments according to RECIST 1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Complete Response (CR) = Disappearance of all target lesions and non-target lesions, Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions with no progression in non-target lesions and no new lesions.
Time Frame: Evaluated every 6 - 9 weeks following treatment initiation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine | CDX-011
Number analyzed (Participants) | 21 | 46
months | 4.2 [2.7 to 5.6] | 2.8 [2.3 to 5.5]

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the number of months from randomization to the date of death due to any cause.
Time Frame: During treatment and 3 months from end of treatment through end of study or approximately up to 5 years.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CDX-011: CDX-011 administered as on Day 1 of each 21 day cycle until disease progression, discontinuation due to toxicity, withdrawal of consent, or end of study.
Arm/Group | Capecitabine | CDX-011
Number analyzed (Participants) | 109 | 218
months | 8.7 [6.9 to 10.8] | 8.9 [7.9 to 10.5]
Statistical Analysis 1: Comparison: Capecitabine vs CDX-011; Test type: Superiority; p = 0.726, Log Rank; Stratified log rank

5. Secondary Outcome: Adverse Events (AE)
Description: The percentage of patients experiencing one or more adverse events will be summarized by treatment arm, relationship to study drug, and severity.
Time Frame: Usually following at least 1 cycle of study treatment (1 dose of CDX-011 or capecitabine and until discontinuation of follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine | CDX-011
Number analyzed (Participants) | 92 | 213
Participants
  Patients with at least 1 AE | 92 | 211
  Patients with at least 1 treatment related AE | 84 | 204
  Patients with Grade 1 treatment related AE | 7 | 7
  Patients with Grade 2 treatment related AE | 33 | 54
  Patients with Grade 3 treatment related AE | 44 | 114
  Patients with Grade 4 treatment related AE | 8 | 32
  Patients with Grade 5 treatment related AE | 0 | 4

6. Secondary Outcome: Pharmacokinetics (PK)
Description: Concentration of the antibody drug conjugate (ADC), total antibody (TA) and free MMAE will be determined.
Time Frame: Following 1 dose of CDX-011.
Population: Samples were obtained from 201 of 213 patients treated with CDX-011. A partial analysis provided below results. Additional analyses were not completed. Results should be interpreted with caution.
Measure: Mean (Full Range); unit: ug/ml
Arm/Group | CDX-011
Number analyzed (Participants) | 201
ug/ml
  Cycle 1 post infusion ADC levels: number analyzed (Participants) | 12
  Cycle 1 post infusion ADC levels | 58.6 [38.8 to 98.3]
  Cycle 1 post infusion TA levels: number analyzed (Participants) | 163
  Cycle 1 post infusion TA levels | 49.4 [21.4 to 127.4]
  Cycle 1 post infusion MMAE levels: number analyzed (Participants) | 47
  Cycle 1 post infusion MMAE levels | 0.0015 [0.0004 to 0.005]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time a subject took their first dose of study treatment (CDX-011 or Capecitabine) through (whichever occurs first) either a) 28 calendar days after the last administration of study treatment, or b) initiation of alternate anticancer therapy.
Arm/Group | Capecitabine | CDX-011
All-Cause Mortality (participants affected / at risk) | 65/92 | 134/213
Serious Adverse Events (participants affected / at risk) | 19/92 | 71/213
Other Adverse Events (participants affected / at risk) | 91/92 | 211/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=92) | CDX-011 (N=213)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 6
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 8
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 4 | 7
Asthenia (General disorders) | 0 | 1
Axillary pain (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 0 | 2
Influenza like illness (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pain (General disorders) | 0 | 3
Polyserositis (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 7
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Bacterascites (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 1
Chest wall abcess (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 5
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 5
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma compliaction (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Erthyema (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=92) | CDX-011 (N=213)
Anaemia (Blood and lymphatic system disorders) | 9 | 33
Neutropenia (Blood and lymphatic system disorders) | 5 | 49
Abdominal distension (Gastrointestinal disorders) | 3 | 12
Abdominal pain (Gastrointestinal disorders) | 16 | 22
Abdominal pain upper (Gastrointestinal disorders) | 6 | 17
Constipation (Gastrointestinal disorders) | 13 | 61
Diarrhoea (Gastrointestinal disorders) | 44 | 55
Dyspepsia (Gastrointestinal disorders) | 4 | 22
Dysphagia (Gastrointestinal disorders) | 0 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 16
Nausea (Gastrointestinal disorders) | 39 | 91
Oral pain (Gastrointestinal disorders) | 2 | 11
Stomatitis (Gastrointestinal disorders) | 24 | 37
Vomiting (Gastrointestinal disorders) | 17 | 46
Asthenia (General disorders) | 5 | 14
Chills (General disorders) | 4 | 14
Fatigue (General disorders) | 37 | 101
Non-cardiac chest pain (General disorders) | 5 | 4
Oedema peripheral (General disorders) | 10 | 13
Pain (General disorders) | 4 | 21
Pyrexia (General disorders) | 12 | 37
Oral candidiasis (Infections and infestations) | 1 | 18
Urinary tract infection (Infections and infestations) | 3 | 18
Alanine aminotransferase increased (Investigations) | 3 | 23
Asparate aminotransferase increased (Investigations) | 6 | 25
Blood alkaline phosphotase increased (Investigations) | 2 | 18
Lymphocyte count decreased (Investigations) | 3 | 12
Neutrophil count decreased (Investigations) | 1 | 38
Weight decreased (Investigations) | 5 | 37
White blood cell count decreased (Investigations) | 2 | 24
Decreased appetite (Metabolism and nutrition disorders) | 17 | 63
Dehydration (Metabolism and nutrition disorders) | 6 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 24
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 38
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 24
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 25
Dizziness (Nervous system disorders) | 4 | 19
Dysgeusia (Nervous system disorders) | 2 | 23
Headache (Nervous system disorders) | 5 | 39
Neuropathy peripheral (Nervous system disorders) | 4 | 28
Paraesthesia (Nervous system disorders) | 5 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 47
Anxiety (Psychiatric disorders) | 5 | 15
Insomnia (Psychiatric disorders) | 6 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 88
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 8
Palmar-plantar erythrodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 40 | 10
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 69
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 | 12
Rash (Skin and subcutaneous tissue disorders) | 3 | 29
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 15
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 11
Rash macular-papular (Skin and subcutaneous tissue disorders) | 5 | 40
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 18
Skin hyerppigmentation (Skin and subcutaneous tissue disorders) | 3 | 19
Dry mouth (Gastrointestinal disorders) | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT01997333/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT01997333/SAP_001.pdf